CLINICAL TRIAL: NCT02669420
Title: Intra Uterine Extra Amniotic (200 μg ) Versus Vaginal (200 μg) Misoprostol for Second Trimester Pregnancy Termination: Randomized Controlled Trial
Brief Title: Misoprostol for Second Trimester Pregnancy Termination
Acronym: MIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, abo bakr mitwally, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 220
Record Dates: First submitted 2016-01-23; First posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Intra Uterine Fetal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- extra amniotic misoprostol (Experimental): misoprostol dissolved in warm saline , become dissolute misoprostol saline solution(200 microgram every 4 hours)
  Interventions: Procedure: termination of second trimester pregnancy
- vaginal misoprostol (Experimental): misoprostol tablet soaked with distilled water and inserted in the posterior fornix of the vagina( 200 microgram every 4 hours)
  Interventions: Procedure: termination of second trimester pregnancy

INTERVENTIONS:
Procedure: termination of second trimester pregnancy — Intra uterine extra amniotic (200 μg ) versus Vaginal (200 μg) Misoprostol for Second Trimester Pregnancy Termination. Randomized controlled trial

SUMMARY:
The majority of second-trimester pregnancy termination performed in the United States are performed surgically by dilation and evacuation. The frequency of induction of abortion increases as gestational age advances. In the late second trimester and early third trimester, induction is the primary method of termination in cases of fetal abnormalities. In many other countries, however, induction is the primary method of abortion throughout the second trimester

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy 13-24 weeks.
* Women with indication for termination of the pregnancy due to intra uterine fetal death

Exclusion Criteria:-Pregnancy before 13 weeks.

* Pregnancy beyond 24 weeks.
* Women with scared uterus.
* Known hypersensitivity for misoprostol.
* Refusal of the woman to participate.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
mean duration from the initial misoprostol dose until complete fetal expulsion | 24 hours

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ghosh J, Papadopoulou A, Devall AJ, Jeffery HC, Beeson LE, Do V, Price MJ, Tobias A, Tuncalp O, Lavelanet A, Gulmezoglu AM, Coomarasamy A, Gallos ID. Methods for managing miscarriage: a network meta-analysis. Cochrane Database Syst Rev. 2021 Jun 1;6(6):CD012602. doi: 10.1002/14651858.CD012602.pub2. PMID 34061352